CLINICAL TRIAL: NCT06786325
Title: A Wellcome Leap for the Opioid Crisis: Can the 5HT2A Agonist Psilocybin Improve Brain, Behavioral, and Clinical Outcomes in Opioid Use Disorder (OUD)?
Brief Title: Wellcome Leap Psilocybin for OUD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anna Rose Childress, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Anna Rose Childress, Ph.D., Research Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 856720
Record Dates: First submitted 2024-12-16; First posted 2025-01-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose Psilocybin (Experimental): 25 mg PEX010 capsule, single dose
  Interventions: Drug: Psilocybin
- Low Dose Psilocybin (Active Comparator): 1 mg PEX010 capsule, single dose
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — PEX010 is the Psilocybin produced by Filament
  Other Names: PEX010

SUMMARY:
Investigators will recruit 36 individuals on MAT for OUD for a double-blind, placebo-controlled design to determine whether PEX010 (25-mg/d) shows preliminary efficacy on neural correlates of neurocognition and on clinical outcomes. Participants will be randomized to either (single dose) 25-mg (PEX010-25 group) or 1-mg (PPEX010-1 group) PEX010 in a 2:1 ratio. Brain and behavioral testing sessions will precede Psilocybin (PSI) dosing day by 24-48 hours and will follow PSI dosing by 1 week. After an initial 6 phases, participants will come into the lab to submit a urine screen 2x/week and to complete a short survey in order to collect data on drug use, MAT adherence, and mental health symptoms. The investigators hypothesize the PEX010-25 (vs. PEX010-1) group will have better clinical outcomes (e.g., lower average percent positive urine drug screens, more late relapses, higher MAT adherence). There are research follow ups every three months out to one year post dose.

DETAILED DESCRIPTION:
The Opioid Crisis: Currently in its third wave, the opioid epidemic involves the prevalence of lethal levels of fentanyl in drugs, leading to a surge in opioid-related deaths. Reports indicate a record-breaking number of over 107,000 drug-related overdose deaths in 2021-2022, with opioids contributing to more than 75% of these fatalities. Beyond fatal overdoses, nearly 1 million non-fatal overdoses occurred in 2017, carrying significant, long-lasting consequences. Those who experience non-fatal overdoses are more prone to subsequent overdoses and have a higher likelihood of death within a year, primarily due to drug-related issues. The escalating cases of opioid use disorder (OUD) emphasize the critical need for innovative treatments to address the associated challenges, including neurocognitive difficulties and poor clinical outcomes. While medication-assisted treatment (MAT) like methadone or buprenorphine effectively alleviates withdrawal symptoms and reduces overdose risk, illicit drug use persists, and non-adherence to MAT remains a challenge. The opioid overdose crisis demands urgent attention and necessitates the development of treatments capable of making a significant impact.

Psilocybin: In response to the need for improved treatments, there's a growing interest in psychedelic-assisted treatment (PAT), particularly involving psilocybin (PSI). Clinical trials support the use of PAT in controlled medical contexts, with 105 trials registered in the past 20 years covering various mental health and other conditions. PSI (at single doses in the proposed range) has shown preliminary promise for depression, alcohol use disorder, and tobacco-use disorder. However, its potential benefits for OUD remain unknown. This proposal aims to determine whether PSI enhances critical OUD clinical outcomes, such as relapse, overdose, and MAT adherence. Importantly, the investigators will test how PSI produces its benefits through its impact on brain and bio-behavioral targets, thus linking potential biomarkers to clinical outcomes.

Cognitive Flexibility: The ability to change thoughts, emotions, and behaviors in response to changes in circumstance (to "flex") has strong survival value. When the brain cannot "flex", one can experience a range of mishaps, from small (turning left rather than right 'out of habit') to much larger ones. Being 'stuck' is a problem that appears in many disorders. For example, individuals with depression may get 'stuck' in dark ruminating thoughts; individuals with OCD may get 'stuck' in repetitive thoughts and behaviors; people with substance use disorders get 'stuck' over-responding to drug reward signals and pursue the drug despite negative consequences. Recent research shows that PSI facilitates intermediate and long-term improvements in cognitive flexibility, raising the hope that it can 're-set' the brain and enable new thoughts, emotions, and behaviors. Cognitive flexibility is often measured by tasks that quantify how successfully one can shift between changing mental rules to complete a task. Using such tasks, there is evidence of cognitive flexibility deficits in people with OUD, but research has not specifically examined the impact of improved cognitive flexibility on OUD clinical outcomes. To date, one study showed that neurocognitive training in executive function (EF), including cognitive flexibility, is associated with reduced opioid use, while a non-OUD study found that higher baseline cognitive flexibility was related to better substance use treatment retention. This proposal will be the first to test whether putative PSI-related improvements in cognitive flexibility will lead to more favorable OUD clinical outcomes.

Other Executive Functions: Importantly, cognitive flexibility is a complex capability that depends on the integrated action of several other basic executive functions (EFs): attention, working memory, and inhibition of thoughts, feelings, or actions. Further, each of these basic EFs, together with cognitive flexibility, are needed for effective and efficient planning and decision-making. Individuals who use drugs demonstrate impairment in a variety of these fundamental EFs. In OUD populations, deficits are evident across most EF domains, including working memory, attention, inhibition, and decision-making, which may relate to or underly their cognitive inflexibility. Studies have found that performance on EF tasks (and the neural underpinnings of EF in the prefrontal cortex [PFC]) indeed correlate with clinical outcomes such as treatment non-adherence (e.g., working memory) and drug use/relapse (e.g., poor inhibition) in substance-use disorders generally, and with reduced abstinence in OUD. Whether these multiple EF deficits predate, or even predispose, drug use - they are likely compounded by drug exposure, including non-fatal opioid overdoses that produce hypoxic-related brain injuries, leading to further neurocognitive deficits. In sum, there is good preliminary evidence for deficits in the several component EFs underlying cognitive flexibility in OUD. By measuring these separately, the current proposal will be able to determine which of these targets are most impacted by PSI, and their relative importance for outcome prediction.

What's "special" about psilocybin? PSI has likely been in use by humans for millennia, originally as a religious or spiritual agent due to its dramatic subjective effects, including hallucinations and mystical experiences. However, scientists have more recently understood that some of the effects - such as increased sense of connectedness, openness, and change in perspective - can produce long-lasting change and improved mental health. Indeed, psychometric instruments capturing non-ordinary states of consciousness and psychological constructs have reliably predicted clinical treatment outcomes, including substance use disorder outcomes. Some theorists have proposed that these dramatic drug effects may reflect a profound initial 'loosening' of top-down control over limbic and sensory regions, resulting in improved flexibility and adaptive behavior. Though the current proposal will not be able to test all features of this hypothesis, the investigators will capture the special acute phenomenology of the drug state and test for the fundamental feature of flexibility. Further, the investigators will determine the relative role of the basic EF components of flexibility and test the importance of all these factors (alone and in combination) for obtaining clinical benefit from the drug. This study will provide a critical foundation for understanding the potential of 5HT2A agonists in OUD, with treatment implications for several other disorders where cognitive inflexibility, 'getting stuck', is a core feature.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document voluntarily signed and dated by the subject.
* Voluntary enrollment in the residential addiction treatment facility
* Intention on residing within residential addiction treatment facility for the duration of the Pre/Post PSI dosing period.
* Either 1) have a confirmed prescription for BUP-NX in a drug monitoring program database, have been on a stable dose of BUP-NX for at least one week, and plan to continue taking BUP-NX for at least 12 weeks or 2) have received an injection of Sublocade® within the past month, or 3) are currently on methadone maintenance therapy and on a consistent dose for at least a week. Subject must provide a urine that is buprenorphine-positive (for subjects taking buprenorphine) or methadone-positive (for subjects taking methadone), during screening.
* Physically healthy males and females, aged 18-60 years old, who meet criteria for opioid use disorder (based on DSM-5 criteria) as their primary diagnosis and are voluntarily seeking treatment.
* Females must be non-pregnant and non-lactating. Additionally, for females with childbearing potential (i.e., have not undergone sterilization via hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, or at least 1 year post-menopausal) participants must agree to use an acceptable form of contraception (e.g. abstinence, intrauterine device, hormonal injection, hormonal implant, hormonal patch/ring/pill, condoms (male or female), etc.) during study participation and to continue its use for the duration of the study
* Subject must read at or above eighth grade level and speak, understand, and write in English.
* IQ score of greater than or equal to 80.

Exclusion Criteria:

* Participation in clinical trial and receipt of investigational drug(s) during 30 days prior to the research study, except as explicitly approved by the Principal Investigator.
* Currently meets DSM-5 criteria for moderate to severe substance use disorder for any substance other than cocaine, alcohol, marijuana or nicotine as determined by the semi-structured interview. Patients with comorbid Alcohol Use Disorder will be accepted if their alcohol use disorder is not severe enough to require a medicated alcohol detoxiﬁcation.
* Meets current or lifetime DSM-5 criteria for schizophrenia or any psychotic disorder, or organic mental disorder or has a first-degree family history of these disorders
* Meets current DSM-5 criteria for bipolar disorder
* Meets current DSM-5 criteria for severe Major Depressive Disorder (mild and moderate MDD as well as in stable remission are allowed if no suicidal risk and no ongoing antidepressant therapy).
* Current or past significant trauma exposure with elevated Post-Traumatic Stress symptoms at the discretion of the PI.
* Presence of any another psychiatric disorder that in the opinion of the PI will interfere with completion of the study or place the patient at heightened risk through participation in the study.
* Current or past month active suicidal ideations or lifetime history of serious suicidal attempt.
* Has evidence of a history of signiﬁcant active hepatitis, signiﬁcant hepatocellular injury as evidenced by elevated bilirubin levels (greater than 1.3), or, pulmonary, endocrine, cardiovascular, renal (creatinine clearance less than or equal to 60ml/min) or gastrointestinal disease, or current HIV infection, and/or clinically signiﬁcant levels (over 3.5x upper limit of normal) of aspartate aminotransferase (AST), and serumalanine aminotransferase (ALT).
* History of serious head trauma or injury causing loss of consciousness that lasted more than 3 minutes and/or associated with skull fracture or intracranial bleeding or abnormal MRI.
* Seizure disorder or history of seizures not related to drug or alcohol withdrawal (excluding childhood febrile seizure).
* Presence of magnetically active prosthetics, plates, pins, broken needles, permanent retainer, bullets, etc. in patient's body (unless a radiologist conﬁrms that its presence is unproblematic). An x-ray may be obtained to determine eligibility.
* Claustrophobia or other medical condition that disables the participant from lying in the MRI for approximately 60 minutes.
* Non-removable skin patches, at discretion of PI.
* Has received medication that could interact adversely with psilocybin within the time of administration of study agent based on the Medical Director's guidance.
* Needs treatment with any psychoactive (e.g., anti-depressants) medications (with the exception of Benadryl used sparingly, if necessary, for sleep).
* *Have the following cardiovascular conditions:

  * coronary artery disease, congenital long QT syndrome (prior diagnosis), cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction (prior diagnosis);
  * tachycardia (deﬁned as heart rate greater than 100 beats per minute);
  * a clinically signiﬁcant Screening ECG abnormality (e.g., atrial ﬁbrillation); Note: A QTcF interval greater than 450 milliseconds is considered a clinically signiﬁcant ECG abnormality
  * artiﬁcial heart valve;
  * any other signiﬁcant current or history of cardiovascular condition, based on the clinical judgment of Medical Director, that would make a participant unsuitable for the study.
* *At Screening or Baseline have elevated blood pressure as deﬁned as:

  * Screening blood pressure SBP greater than135 mmHg or DBP greater than 85 mmHg on three separate readings; or
  * Baseline blood pressure SBP greater than140 mmHg or DBP greater than 90 mmHg on three separate readings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percent of patients in each arm having urine drug screens positive for opioids | weeks 1 through 8 (outcomes phase)
  Urine drug screen (UDS), percent positive illicit opioids (e.g., fentanyl) during the 8-week outpatient phase, calculated by taking number of positive detections by total number of opportunities to submit UDS (2 per week for 8 weeks equals 16 opportunities). This variable will be a single, continuous variable measured as a percentage. As well as self-reported drug use via TLFB.
MAT adherence as recorded by self report and corroborated POC UDS tests during the twicely weekly outcomes phase visits | weeks 1 through 8 outpatient phase
  Self-reported use of prescribed MAT for OUD via TLFB; MAT metabolites (e.g., buprenorphine, methadone) will be detectable in twice-weekly urine drug screens, calculated by taking number of positive detections of MAT metabolites divided by the number of opportunities to submit a UDS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No